CLINICAL TRIAL: NCT00438282
Title: Age 6 Test of Home Visits by Nurses vs Paraprofessionals
Acronym: DenverY06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Colorado Trust (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 00-0036; R01MH062485 (NIH); NCT00053664 (obsolete NCT alias)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-02

CONDITIONS: Child Rearing; Risk Reduction Behavior; Reproductive Behavior
Keywords: nurse; home visits; pregnancy; welfare; child development
MeSH Terms: conditions — Risk Reduction Behavior; Reproductive Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Control group
- 2 (Experimental): Paraprofessional home visits
  Interventions: Behavioral: home visitation
- 3 (Experimental): Nurse home visitation
  Interventions: Behavioral: home visitation

INTERVENTIONS:
Behavioral: home visitation — Home visitation from midway through pregnancy until child age 2. Group 2 is visitation by Paraprofessionals; group 3 is home visitation by Nurses.
  Arms: 2; 3

SUMMARY:
To examine the impact of prenatal and infancy home visiting by paraprofessionals and by nurses from child age 2 through 6.

DETAILED DESCRIPTION:
This project supports an age-six assessment of 669 children and their families who were enrolled in a randomized trail that compared prenatal and infancy home visiting by nurses versus paraprofessionals. Both groups of visitors in each study employed essentially the same program model. The program model has proven to be effective using nurses when focused on European-American and African Americans in earlier trails conducted over the past 20 years. Paraprofessional visitors in the current trail share many of the social characteristics of the families they visited. The current study also allows us to examine the extent to which these different visitor types produce effects with Mexican Americans that are similar to those achieved with European-Americans and African Americans in previous trails of this program using nurse home visitors. The sample is composed of low-income women who had no previous live births and who were substantially ethnic minorities (46 percent Mexican American, 16 percent African American, and 3 percent Native American/Asian), unmarried (87 percent), and less than 19 years of age (58 percent) at the time of registration during pregnancy.

In earlier phases of assessment, the nurse-visitor program was found to reduce women's use of tobacco during pregnancy; to improve the home environments and quality of care that mothers provided to their children; to improve the language and mental development of children born to mothers with low psychological resources (where psychological resources were defined as high rates of mental disorder symptoms, limited intellectual functioning, and little belief in their control over their life circumstances); and to improve maternal life-course, as reflected in fewer subsequent pregnancies and increases in employment. The paraprofessional program produced smaller, mostly non-significant and inconsistent effects while the program was in operation, but recent evidence from a 4-year follow up of the sample now suggests that paraprofessional program effects on parental caregiving and child development may be increasing as the children mature. The current proposal seeks support to determine whether the beneficial effects of the nurse home visiting program endure through the children's completion of kindergarten at age six, and whether beneficial effects emerge at this later time period for families visited by paraprofessionals.

ELIGIBILITY:
Inclusion Criteria:

* Women were recruited from 21 antepartum clinics serving low-income women in Denver if they had no previous live births and either qualified for Medicaid or had no private insurance.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2001-03; Primary Completion 2005-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
increased interval between the birth of the first and second child; | When first child is 6
increased cohabitation with the biological father of the child and the involvement of a supportive male partner; | When first child is 6
increase parents' competent care of their children, as reflected in greater involvement and monitoring of their children's behavior, more consistent discipline, and greater investment in their children's educational achievement. | When first child is 6
children's behavior problems and expressions of dysregulated aggressive and violent themes in their response to the MacArthur Story Stem Battery | When child is 6
children's compromised executive functions, language and intellectual skills | When child is 6

CONTACTS AND LOCATIONS:
Overall Officials: David L Olds, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] Olds DL, Robinson J, Pettitt L, Luckey DW, Holmberg J, Ng RK, Isacks K, Sheff K, Henderson CR Jr. Effects of home visits by paraprofessionals and by nurses: age 4 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1560-8. doi: 10.1542/peds.2004-0961. PMID 15574615
- [Background] Olds DL, Robinson J, O'Brien R, Luckey DW, Pettitt LM, Henderson CR Jr, Ng RK, Sheff KL, Korfmacher J, Hiatt S, Talmi A. Home visiting by paraprofessionals and by nurses: a randomized, controlled trial. Pediatrics. 2002 Sep;110(3):486-96. doi: 10.1542/peds.110.3.486. PMID 12205249
- [Derived] Olds DL, Holmberg JR, Donelan-McCall N, Luckey DW, Knudtson MD, Robinson J. Effects of home visits by paraprofessionals and by nurses on children: follow-up of a randomized trial at ages 6 and 9 years. JAMA Pediatr. 2014 Feb;168(2):114-21. doi: 10.1001/jamapediatrics.2013.3817. PMID 24296904